CLINICAL TRIAL: NCT07084012
Title: A Phase IIa Randomized, Blinded, Placebo-Controlled Clinical Trial to Evaluate the Efficacy and Safety of Intravenous Infusion of Human Umbilical Cord Mesenchymal Stem Cells (hUC-MSCs) in the Treatment of Acute Ischemic Stroke (AIS)
Brief Title: A Phase IIa Clinical Trial to Evaluate the Efficacy and Safety of Intravenous Infusion of hUC-MSCs in Patients With AIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Wingor Biotechnology Co., Ltd. (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WG103-AIS-Ⅱa
Record Dates: First submitted 2025-07-08; First posted 2025-07-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke AIS
Keywords: hUC-MSCs; AIS,; Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Subjects receive one infusion of hUC-MSCs infusions.
  Interventions: Drug: hUC-MSCs treatment (high dose)
- Group 2 (Experimental): Subjects receive three infusions of hUC-MSCs.
  Interventions: Drug: hUC-MSCs treatment (low dose)
- Placebo Control Group (Placebo Comparator): Subjects receive three infusions of cell medium placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hUC-MSCs treatment (high dose) — 2.0×10^8 cells per infusion, single administration on D0. Infusion of cell medium placebo on Day 7 (±2 days), and Day 14 (±2 days).
  Other Names: hUC-MSCs injection
  Arms: Group 1
Drug: hUC-MSCs treatment (low dose) — 1.0×10^8 cells per infusion, 3 administrations, on Day 0, Day 7 (±2 days), and Day 14 (±2 days)
  Other Names: hUC-MSCs injection
  Arms: Group 2
Drug: Placebo — Cell medium, 3 administrations, on Day 0, Day 7 (±2 days), and Day 14 (±2 days)
  Arms: Placebo Control Group

SUMMARY:
This is a Phase IIa clinical trial with a three-arm design that utilizes randomization, double-blinding, and placebo control. The primary objective of this study is to evaluate the efficacy of single and multiple intravenous infusions of hUC-MSCs injection in patients with AIS. The secondary objective is to assess the safety and tolerability of single and multiple intravenous infusions of hUC-MSCs injection in patients with AIS. The exploratory objective is to investigate the pharmacokinetic and pharmacodynamic characteristics of hUC-MSCs injection in patients with AIS.

DETAILED DESCRIPTION:
Stroke is a disease with high incidence, disability rate, and mortality rate, ranking as the second leading cause of death globally and the leading cause in China. Acute ischemic stroke (AIS) accounts for approximately 60%-80% of all strokes. The most effective treatments for AIS are revascularization therapies within the time window, including intravenous thrombolysis with tissue plasminogen activator (t-PA) and mechanical thrombectomy. Although t-PA thrombolysis is effective, it can cause reperfusion injury, exacerbating a series of inflammatory damages. Additionally, the success rate of thrombolysis and thrombectomy is closely related to the onset time. The time window within 4.5 hours or 6 hours is considered effective for rescuing the ischemic penumbra, and only a minority of AIS patients can receive thrombolytic therapy. Some patients have contraindications to thrombolysis, and endovascular treatment is only suitable for large vessel occlusion. Furthermore, in China, low public awareness of early disease recognition, insufficient prehospital emergency capabilities, in-hospital emergency delays, and other factors lead to delayed AIS treatment and a low thrombolysis rate.

Studies have shown that mesenchymal stem cells can reduce the infarct area and alleviate blood-brain barrier damage by regulating the microenvironment of damaged brain tissue, alleviating inflammatory responses, and promoting angiogenesis, neurogenesis, and neurovascular repair. This study aims to evaluate the efficacy, safety, and tolerance of single and multiple intravenous infusions of hUC-MSCs injection in the treatment of AIS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years, inclusive, regardless of gender.
2. Diagnosis of acute ischemic stroke (AIS).
3. Onset time ≤ 72 hours.
4. Anterior circulation cerebral infarction.
5. Modified Rankin Scale (mRS) score ≤ 1 before the onset of this stroke.
6. National Institutes of Health Stroke Scale (NIHSS) score between 8 and 20 (inclusive) at screening, and NIHSS item 1a (level of consciousness) score ≤ 1.
7. The subject or their legal guardian has signed the informed consent form.

Exclusion Criteria:

1. Planned or already undergone thrombolysis or thrombectomy for this stroke.
2. History of epilepsy (excluding secondary epilepsy that does not currently require medication), Parkinson's disease, Alzheimer's disease, severe depression, or other diseases that the investigator deems would affect the subject's participation in the trial or the assessment of efficacy.
3. Presence of intracranial hemorrhagic disease (e.g., intracerebral hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural/epidural hematoma, etc.). If only petechial bleeding is present, the investigator may determine whether the subject is suitable for inclusion in the study.
4. Computed tomography (CT) or magnetic resonance imaging (MRI) of the head showing a large ischemic area in the middle cerebral artery territory or midline shift greater than 1 cm on head CT/MRI, and the investigator assesses a high likelihood of surgical intervention or poor prognosis.
5. Presence of brain tumor or history of malignancy.
6. Liver or kidney insufficiency during the screening period: Aspartate aminotransferase (AST) > 2.5 × upper limit of normal, alanine aminotransferase (ALT) > 2.5 × upper limit of normal, estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m².
7. History of severe cardiovascular disease, which the investigator deems unsuitable for participation in this clinical trial.
8. Severe infection, including sepsis, septic shock, severe pneumonia, etc.
9. Systemic corticosteroid ( > 10 mg/day prednisone equivalent) or immunosuppressive drug treatment within 14 days before receiving the investigational drug or during the trial.
10. History of alcohol abuse within the past year (defined as an average of more than 2 units per day (1 unit = 10 mL ethanol, i.e., 1 unit = 200 mL of 5% alcohol beer or 25 mL of 40% alcohol spirits or 85 mL of 12% alcohol wine).
11. Pregnant or breastfeeding women; or unwillingness to use reliable contraception (e.g., condoms) throughout the study period, or plans to donate sperm or eggs, or have plans for pregnancy.
12. Participation in an interventional clinical trial within the past 3 months, or receipt of other cell therapy (excluding blood transfusion).
13. Other situations in which the investigator deems the patient unsuitable for participation in this study (including but not limited to non-compliance with the principle of patient benefit, poor patient compliance, unacceptable laboratory abnormalities, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with an mRS score of 0-2 at different follow-up visits after treatment. | 360 days
  Evaluate each patient's modified Rankin Scale (mRS) score, with a total score ranging from 0 to 6, where a higher score indicates a poorer outcome. Determine the proportion of patients with an mRS score of 0-2 at different follow-ups after treatment.
The proportion of subjects with an NIHSS improvement of ≥4 points at different follow-up visits after treatment | 90 days
  Evaluate each patient's National Institutes of Health Stroke Scale (NIHSS) score at different follow-up time points after treatment.
  The NIHSS score ranges from 0 to 42, with higher scores indicating more severe neurological impairment.
  Determine the proportion of subjects with an improvement of ≥4 points in their NIHSS score.
Changes in NIHSS score from baseline at different follow-up visits after treatment | 90 days
  Evaluate each patient's National Institutes of Health Stroke Scale (NIHSS) score before treatment and at different follow-up time points after treatment.
  The NIHSS score ranges from 0 to 42, with higher scores indicating more severe neurological impairment.
  Determine the changes in NIHSS scores relative to the baseline.
Trends in the distribution of mRS scores (0-6) at different follow-up visits after treatment | 360 days
  Evaluate the modified Rankin Scale (mRS) score for each patient, with a total score ranging from 0 to 6, where a higher score indicates a poorer outcome. Determine the distribution trend of mRS scores (0-6) at different follow-up visits after treatment.
The proportion of subjects with a Barthel Index (BI) score of ≥95 at different follow-up visits after treatment | 360 days
  Evaluate the Barthel Index of Activities of Daily Living (BI) score for each patient, which ranges from 0 to 100, with higher scores indicating better independence and less dependence of the patient.
  Determine the proportion of subjects with a BI score of ≥95 at different follow-up visits after treatment.
Changes in Fugl-Meyer Motor Function Assessment Scale score from baseline at different follow-up visits after treatment | 360 days
  Evaluate the Fugl-Meyer Motor Function Assessment Scale score for each patient before and after treatment.
  The scale consists of 50 items, with a maximum total score of 100, where a higher score indicates a better outcome.
  Determine the change in Fugl-Meyer Motor Function Assessment Scale score from baseline at different follow-up visits after treatment.

SECONDARY OUTCOMES:
Adverse Events | 360 days
  Adverse Events: Including AEs , SAEs , any AE leading to discontinuation of treatment, any adverse reaction occurring in subjects within 180 days, and neurologic deterioration related to the drug.
All-cause mortality rate | 360 days
  All-cause mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No